CLINICAL TRIAL: NCT01318798
Title: Development and Validation of an Enhanced Prediction Score for Post-operative Acute Renal Failure Following Liver Resection
Brief Title: Development and Validation of an Enhanced Prediction Score for Postoperative Acute Renal Failure After Liver Resection
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Ksenija Slankamenac, Md PhD, University of Zurich
Other Study IDs: StV 33-2009
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Acute Renal Failure
Keywords: Development; Pre- and intra-operative predictors; Acute renal failure; Liver Surgery; Prediction score; Validation; Clinical consequences; Decision curve analysis; predictors of acute renal failure after liver resection
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with post-operative ARF: Patients developing acute renal failure (ARF) following liver surgery
  ARF was defined according to the RIFLE criteria as an absolute increase in serum-creatinine of more than 0.3 mg/dl above baseline, or an increase of more than 1.5 times the pre-operative baseline value within 48 hours after surgery, or a reduction of urinary output less than 0.5 ml/kg/h for at least 6 hrs.
- Patients without post-operative ARF: Patients with normal kidney function (without acute renal failure (ARF)) following liver surgery

SUMMARY:
Post-operative acute renal failure is a severe post-operative complication and is associated with high mortality. The enhanced prediction score, including pre-as well as intra-operative predictors accurately predicted ARF following hepatic surgery. This prediction score allows early identification of patients at high risk of ARF and may support decision-making for protective kidney treatment.

DETAILED DESCRIPTION:
To enhance and validate an already pre-existing score accurately predicting post-operative acute renal failure (ARF) after hepatic surgery

We will enhance a pre-existing score predicting ARF based on pre-operative as well as intra-operative predictors.

Development process: we will identify the strongest predictors of ARF in a multivariable logistic regression model followed by a stepwise backward logistic regression analysis and bootstrapping.

Validation process: we will perform an internal validation by calibrating the prediction model as well as by k-fold cross validation (c statistics) and bootstrapping. Additionally, we will calculate the discrimination by the area under the curve (AUC).

Decision curve analysis: Furthermore we will perform a decision curve analysis to evaluate the clinical consequences of both prediction scores whether a patient with increased ARF risk would post-operative benefit of a treatment on the ICU.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* scheduled for liver surgery
* benign as well as malignant diseases

Exclusion Criteria:

* liver trauma
* incomplete data sets
* pre-operative chronic renal failure requiring hemodialysis

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included consecutively patients undergoing any type of hepatic surgery for benign as well as malignant diseases between July first, 2002 and October 31, 2007 in a single tertiary care center (Swiss Hepato-Pancreato-Biliary (HPB) Centre, University Hospital of Zurich, Switzerland.
Sampling Method: Probability Sample
Enrollment: 549 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Development of an enhanced prediction score for ARF | within 48 hours post-operative
  Development of an enhanced but still simple and easy applicable score based on pre- and extended by intra-operative risk factors to predict postoperative ARF in patients scheduled for liver resection

SECONDARY OUTCOMES:
Decision curve analysis | within 48 hours post-operative
  Describing a decision making model by performing a decision curve analysis for clinical consequences of the enhanced prediction score and comparing it with the pre-operative prediction score
internal validation of the enhanced prediction score | within 48 hours post-operative
  internal Validation: discrimination, calibration, k-fold cross validation and bootstrapping

CONTACTS AND LOCATIONS:
Overall Officials: Ksenija Slankamenac, med. pract., Principal Investigator — University Hospital Zurich, Visceral and Transplantation Surgery
Locations (1):
- University Hospital of Zurich, Departmente of Visceral and Transplantation Surgery, Zurich, Switzerland

REFERENCES:
- [Result] Slankamenac K, Breitenstein S, Held U, Beck-Schimmer B, Puhan MA, Clavien PA. Development and validation of a prediction score for postoperative acute renal failure following liver resection. Ann Surg. 2009 Nov;250(5):720-8. doi: 10.1097/SLA.0b013e3181bdd840. PMID 19809295